CLINICAL TRIAL: NCT02569476
Title: A Phase 1b Study to Assess Safety, Tolerability and Antitumor Activity of the Combination of BGB 3111 With Obinutuzumab in Subjects With B-Cell Lymphoid Malignancies
Brief Title: BGB 3111 in Combination With Obinutuzumab in Participants With B-Cell Lymphoid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGB-3111_GA101_Study_001
Record Dates: First submitted 2015-09-18; First posted 2015-10-06 (Estimated); Results first posted 2021-11-03 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: B-cell Lymphoid Malignancies
Keywords: BGB-3111; Zanubrutinib; Obinutuzumab; Lymphoma; Leukemia; Therapeutic uses; B-cell
MeSH Terms: conditions — Lymphoma; Leukemia | interventions — zanubrutinib; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Zanubrutinib and Obinutuzumab (Experimental): In the dose-escalation part, dose levels and regimens were evaluated. In the indication-specific expansion cohorts, participants were assigned to different cohorts based on histology type.
  Interventions: Drug: Zanubrutinib; Drug: Obinutuzumab

INTERVENTIONS:
Drug: Zanubrutinib
  Other Names: BGB-3111
Drug: Obinutuzumab

SUMMARY:
This study evaluated the safety and preliminary efficacy of BGB-3111 (zanubrutinib) in combination with obinutuzumab in participants with B-cell lymphoid malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years, able and willing to provide written informed consent and to comply with the study protocol.
* Laboratory parameters as specified below:

  * Hematologic: Platelet count >40x10^9/liter (L) (may be post-transfusion); absolute neutrophil count >1.0x10^9/L (growth factor use is allowed to bring pre-treatment neutrophils to >1.0x10^9 cells/L if marrow infiltration is involved).
  * Hepatic: Total bilirubin <3 x upper limit normal (ULN); and aspartate aminotransferase and alanine transaminase ≤3 x ULN.
  * Renal: Creatinine clearance ≥50 milliliters/minute (as estimated by the Cockcroft Gault equation or as measured by nuclear medicine scan or 24-hour urine collection); participants requiring hemodialysis will be excluded.
* Anticipated survival of at least 6 months.
* Eastern Cooperative Oncology Group performance status of 0 to 2.
* Female participants of childbearing potential and non-sterile males must have agreed to practice at least one of the following methods of birth control with partner(s) throughout the study and for ≥3 months after discontinuing zanubrutinib or ≥18 months following obinutuzumab treatment, whichever was longer: total abstinence from sexual intercourse, double barrier contraception, intra uterine device or hormonal contraceptive initiated at least 3 months prior to first administration of study drug.
* Male participants must have not donated sperm from first study drug administration, until 3 months after zanubrutinib discontinuation or 18 months following obinutuzumab treatment, whichever is longer.

Exclusion Criteria:

* Known central nervous system lymphoma or leukemia.
* Known prolymphocytic leukemia or history of, or currently suspected, Richter's syndrome.
* Uncontrolled autoimmune hemolytic anemia or idiopathic thrombocytopenia purpura.
* History of significant cardiovascular disease.
* Severe or debilitating pulmonary disease.
* History of severe allergic or anaphylactic reactions to monoclonal antibody therapy.
* Prior Bruton tyrosine kinase inhibitor treatment.
* Used medications which were strong cytochrome P450 (CYP) 3A inhibitors and strong CYP3A inducers.
* Vaccination with a live vaccine within 28 days of the initiation of treatment.
* Allogeneic stem cell transplantation within 6 months, or had active graft versus host disease requiring ongoing immunosuppression.
* Receipt of the following treatment prior to first administration of zanubrutinib, corticosteroids given with anti-neoplastic intent within 7 days, chemotherapy or radiotherapy within 3 weeks, monoclonal antibody within 4 weeks.
* Participated in any investigational drug study within 28 days of study entry, or not recovered from non-hematologic toxicity of any prior chemotherapy up to ≤ Grade 1 (except for alopecia).
* History of other active malignancies within 2 years of study entry.
* Major surgery in the past 4 weeks.
* Active symptomatic fungal, bacterial and/or viral infection including evidence of infection with human immunodeficiency virus, human T cell lymphotropic virus seropositive status.
* Inability to comply with the study procedures.
* Pregnant or nursing women.
* Any illness or condition that in the opinion of the investigator may have affected the safety of treatment or evaluation of any study's endpoints.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2016-01-13 (Actual); Primary Completion 2020-09-02 (Actual); Study Completion 2020-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Principal Investigator — BeiGene
Locations (14):
- United States (3):
  - Florida Cancer Specialists Fort Myers, Fort Myers, Florida
  - Florida Cancer Specialists East, West Palm Beach, Florida
  - Tennessee Oncology, Nashville, Tennessee
- Australia (8):
  - St George Hospital, Kogarah, New South Wales
  - Brisbane Clinic For Lymphoma, Greenslopes, Queensland
  - Ashford Cancer Centre Research Northeast, Windsor Gardens, South Australia
  - St Vincents Hospital Melbourne, Fitzroy, Victoria
  - Barwon Health the Geelong Hospital, Geelong, Victoria
  - St Frances Xavier Cabrini Hospital, Malvern, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- South Korea (3):
  - Asan Medical Center, Seoul, Seoul Teugbyeolsi
  - Gangnam Severance Hospital, Yonsei University Health System, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center, Seoul, Seoul Teugbyeolsi

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Tam CS, Quach H, Nicol A, Badoux X, Rose H, Prince HM, Leahy MF, Eek R, Wickham N, Patil SS, Huang J, Prathikanti R, Cohen A, Elstrom R, Reed W, Schneider J, Flinn IW. Zanubrutinib (BGB-3111) plus obinutuzumab in patients with chronic lymphocytic leukemia and follicular lymphoma. Blood Adv. 2020 Oct 13;4(19):4802-4811. doi: 10.1182/bloodadvances.2020002183. PMID 33022066

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 15 study centers in Australia, South Korea, and the United States (US). A total of 119 participants were enrolled in the study and received ≥1 dose of study treatment.
Groups:
- Zanubrutinib and Obinutuzumab: Part 1: Two dose regimens of zanubrutinib (320 milligrams [mg] once daily [QD] and 160 mg twice daily [BID]) in combination with obinutuzumab (dose regimen consistent with the US prescribing information) were evaluated. Part 2: The 2 dose regimens selected from Part 1 (zanubrutinib 320 mg QD and 160 mg BID in combination with obinutuzumab) were investigated in 5 expansion cohorts.
Period: Overall Study
Arm/Group | Zanubrutinib and Obinutuzumab
Started | 119
Completed | 0
Not Completed | 119
Not completed — Roll over to Long-Term Extension Study | 73
Not completed — Death | 33
Not completed — Withdrawal by Subject | 9
Not completed — Progressive disease at study withdrawal and death by end of study | 1
Not completed — Palliative care | 1
Not completed — Transitioned to Long Term Follow Up Study | 1
Not completed — Transitioned to Long Term Extension Study | 1

BASELINE CHARACTERISTICS:
Groups:
- Zanubrutinib and Obinutuzumab: Part 1: Two dose regimens of zanubrutinib (320 mg QD and 160 mg BID) in combination with obinutuzumab (dose regimen consistent with the US prescribing information) were evaluated. Part 2: The 2 dose regimens selected from Part 1 (zanubrutinib 320 mg QD and 160 mg BID in combination with obinutuzumab) were investigated in 5 expansion cohorts.
Arm/Group | Zanubrutinib and Obinutuzumab
Number analyzed (Participants) | 119
Age, Continuous [Median (Full Range); unit: years] | 68 [34 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 78
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 107
  Black or African American | 1
  Asian | 11
  Not Hispanic or Latino | 117
  Hispanic or Latino | 2
Vital Signs [Mean (Standard Deviation); unit: millimeters of mercury]
  Blood Pressure (Systolic) | 124.5 (17.75)
  Blood Pressure (Diastolic) | 71.5 (11.46)
Pulse Rate [Mean (Standard Deviation); unit: beats/minute] | 78.2 (13.86)
Weight [Mean (Standard Deviation); unit: kilograms] | 78.95 (18.004)
Height [Mean (Standard Deviation); unit: centimeters] | 170.92 (9.382)
Body Mass Index [Mean (Standard Deviation); unit: kilograms/squared meter] | 26.876 (4.9513)
Eastern Cooperative Oncology Group [Count of Participants; unit: Participants] — Grade 0: Fully active, able to carry on all pre-disease performance without restriction; Grade 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, eg, light house work, office work; Grade 2: Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours; Grade 0 was considered to be the best outcome.
  Participants
    Grade 0 | 63
    Grade 1 | 48
    Grade 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Part 1 : Number Of Participants Experiencing Adverse Events
Description: An AE was defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product (zanubrutinib in combination with obinutuzumab). An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of the study drug. A serious AE (SAE) was any untoward medical occurrence that, at any dose.
  * resulted in death,
  * was life threatening,
  * required hospitalization or prolongation of existing hospitalization,
  * resulted in disability/incapacity,
  * was a congenital anomaly/birth defect.
Time Frame: Day 1 (first dose) through 4 years and 8 months
Population: Part 1: Safety Analysis Set included all participants who received ≥ 1 dose of zanubrutinib and/or obinutuzumab
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: Zanubrutinib and Obinutuzumab: Part 1: Two dose regimens of zanubrutinib (320 mg QD and 160 mg BID) in combination with obinutuzumab (dose regimen consistent with the US prescribing information) were evaluated.
Arm/Group | Part 1: Zanubrutinib and Obinutuzumab
Number analyzed (Participants) | 12
Participants
  Any TEAE | 12
  SAE | 7

2. Primary Outcome: Part 1: Number Of Participants With Clinical Laboratory Abnormalities
Description: Laboratory results are reported as participants with shifts towards (high directionality) or away (low directionality) from Grade 3 or Higher Toxicity.
Time Frame: Day -28 to -1 (predose) through 4 years and 8 months
Population: The Safety Analysis Set included all participants who received ≥ 1 dose of zanubrutinib and/or obinutuzumab
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: 160 mg BID; Part 1: 320 mg QD: Part 1: Two dose regimens of zanubrutinib (320 mg QD and 160 mg BID) in combination with obinutuzumab (dose regimen consistent with the US prescribing information) were evaluated.
Arm/Group | Part 1: 160 mg BID | Part 1: 320 mg QD
Number analyzed (Participants) | 6 | 6
Participants
  Leukocytes: Low Directionality | 1 | 0
  Lymphocytes: Low Directionality | 1 | 3
  Lymphocytes: High Directionality | 1 | 1
  Neutrophils: Low Directionality | 1 | 3
  Platelets: Low Directionality | 0 | 1
  Phosphate: Low Directionality | 1 | 0
  Urate: High Directionality | 0 | 1

3. Primary Outcome: Part 1: Number Of Deaths
Description: An AE was defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product (zanubrutinib in combination with obinutuzumab). An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study drug. An SAE was any untoward medical occurrence that, at any dose:
  * resulted in death,
  * was life threatening,
  * required hospitalization or prolongation of existing hospitalization,
  * resulted in disability/incapacity,
  * was a congenital anomaly/birth defect.
Time Frame: Day 1 (first dose) through 4 years and 8 months
Population: Part 1: The Safety Analysis Set included all participants who received ≥ 1 dose of zanubrutinib and/or obinutuzumab
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Zanubrutinib and Obinutuzumab
Number analyzed (Participants) | 12
Participants | 0

4. Primary Outcome: Part 1: Number Of Participants Experiencing Dose-limiting Toxicity (DLT)
Description: Dose-limiting toxicities were defined as a toxicity or AE occurring during the DLT assessment period (first 29 days of treatment), which is not clearly attributable to a cause other than zanubrutinib and/or obinutuzumab (such as disease progression, underlying illness, concurrent illness or concomitant medication) and meets one of the following criteria:
  * Grade 3 or 4 drug-related non-hematologic toxicity (excluding Grade 3 nausea, vomiting, hypertension, and asymptomatic laboratory abnormalities),
  * Grade 4 drug-related hematologic toxicity persisting for >14 days,
  * any grade toxicity, which in the judgment of the investigator or Sponsor, required removal of the participant from the study.
Time Frame: Day 1 (first dose) through 4 years and 8 months
Population: Part 1:The Safety Analysis Set included all participants who received ≥ 1 dose of zanubrutinib and/or obinutuzumab
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Zanubrutinib and Obinutuzumab
Number analyzed (Participants) | 12
Participants | 0

5. Primary Outcome: Part 1 and Part 2: Number Of Participants Achieving A Best Response Of Partial Response
Description: Partial response was defined as follows:
  * ≥ 50% reduction of serum IgM from baseline,
  * reduction in lymphadenopathy/splenomegaly (if present at baseline). For response assessments that occurred during cycles where a CT scan was not required, then results from prior scans (up to 12 weeks during the first 48 weeks and up to 24 weeks thereafter) could be carried forward in those participants with extramedullary disease at baseline.
Time Frame: Day 1 (first dose) through 4 years and 8 months
Population: The Safety Analysis Set included all participants who received ≥ 1 dose of zanubrutinib and/or obinutuzumab. The Safety Analysis Set was the primary analysis set for the efficacy and safety analyses.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: Zanubrutinib and Obinutuzumab: Part 1: Two dose regimens of zanubrutinib (320 milligrams [mg] once daily [QD] and 160 mg twice daily [BID]) in combination with obinutuzumab (dose regimen consistent with the US prescribing information) were evaluated. Part 2: The 2 dose regimens selected from Part 1 (zanubrutinib 320 mg QD and 160 mg BID in combination with obinutuzumab) were investigated in 5 expansion cohorts.
Arm/Group | Part 1: Zanubrutinib and Obinutuzumab
Number analyzed (Participants) | 119
Participants | 51

6. Secondary Outcome: Part 1 and Part 2: Number Of Participants Achieving A Best Response Of Complete Response
Description: Complete response was defined as follows:
  * normal serum IgM values,
  * disappearance of monoclonal protein by immunofixation,
  * no histological evidence of bone marrow involvement,
  * complete resolution of lymphadenopathy/splenomegaly (if present at baseline) For response assessments that occurred during cycles where a computed tomography (CT) scan was not required, then results from prior scans (up to 12 weeks during the first 48 weeks and up to 24 weeks thereafter) could be carried forward in those participants with extramedullary disease at baseline.
Time Frame: Day 1 (first dose) through 4 years and 8 months
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Zanubrutinib and Obinutuzumab
Number analyzed (Participants) | 119
Participants | 36

7. Secondary Outcome: Part 1 and Part 2: Progression-free Survival (PFS)
Description: Progression-free survival was defined as time (in months) from the start of treatment with zanubrutinib or obinutuzumab to the first documented disease progression or death due to any cause, whichever occurred first. Results are reported as the median months for each of the B-cell malignancy subtypes: chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL), Waldenström macroglobulinemia (WM), follicular lymphoma (FL), mantle cell lymphoma (MCL), marginal zone lymphoma (MZL), and non-germinal center B-cell-like (GCB) diffuse large B-cell lymphoma (DLBCL).
Time Frame: Day 1 (first dose) through 4 years and 8 months
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1: Zanubrutinib and Obinutuzumab
Number analyzed (Participants) | 119
Months
  WM: number analyzed (Participants) | 7
  WM | 37.13 [6.31 to NA] — NA = Data not estimable due to insufficient number of participants with events
  FL: number analyzed (Participants) | 36
  FL | 24.87 [11.07 to NA] — NA = Data not estimable due to insufficient number of participants with events
  MZL: number analyzed (Participants) | 3
  MZL | 40.25 [8.25 to NA] — NA = Data not estimable due to insufficient number of participants with events
  Non-GCB DLBCL: number analyzed (Participants) | 22
  Non-GCB DLBCL | 2.86 [1.71 to 7.39]
  Total | 40.25 [27.63 to NA] — NA = Data not estimable due to insufficient number of participants with events
  CLL/SLL | NA [44.48 to NA] — NA = Data not estimable due to insufficient number of participants with events

8. Secondary Outcome: Part 1 and Part 2: Duration Of Response (DOR)
Description: Duration of response for responders was defined as the time (in months) from the date of the earliest qualifying response to the date of progressive disease or death due to any cause (whichever occurred earlier). Duration of response was analyzed using the same methods as the analysis for PFS. Responses after initiating new anticancer therapy, roll over to the long-term extension (LTE) study, or the first occurrence of disease progression were not considered in the analysis.
Time Frame: Day 1 (first dose) through 4 years and 8 months
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1: Zanubrutinib and Obinutuzumab
Number analyzed (Participants) | 119
Months
  WM: number analyzed (Participants) | 7
  WM | 35.84 [21.03 to NA] — NA = Data not estimable due to insufficient number of participants with events
  FL: number analyzed (Participants) | 36
  FL | 39.75 [18.63 to NA] — NA = Data not estimable due to insufficient number of participants with events
  Non-GCB DLBCL: number analyzed (Participants) | 22
  Non-GCB DLBCL | 12.75 [2.89 to NA] — NA = Data not estimable due to insufficient number of participants with events
  CLL/SLL | NA [42.02 to NA] — NA = Data not estimable due to insufficient number of participants with events
  MCL | NA [2.73 to NA] — NA = Data not estimable due to insufficient number of participants with events
  MZL | NA [31.80 to NA] — NA = Data not estimable due to insufficient number of participants with events

9. Secondary Outcome: Part 1 and Part 2: Time To Response (TTR)
Description: The TTR for responders was defined as time (in months) from the start of the study treatment to the date of the earliest qualifying response. The TTR was summarized using descriptive statistics. Responses after initiating new anticancer therapy, roll over to the LTE study, or the first occurrence of disease progression were not considered in the analysis of TTR.
Time Frame: Day 1 (first dose) through 4 years and 8 months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Part 1: Zanubrutinib and Obinutuzumab
Number analyzed (Participants) | 119
Months
  CLL/SLL | 3.14 (1.551)
  WM | 2.81 (0.050)
  FL | 3.32 (1.511)
  MCL | 2.77 (0.157)
  MZL | 5.62 (4.042)
  Non-GCB DLBCL | 2.76 (0.297)
  Total | 3.18 (1.487)

10. Secondary Outcome: Part 1 and Part 2: Overall Survival (OS)
Description: Overall survival was defined as the time (in months) from the date of the start of the study treatment to death due to any cause. Participants who were alive before final database lock or discontinuation of the study (discontinued study due to reasons other than death) were censored at their last known alive date on or before database lock.
Time Frame: Day 1 (first dose) through 4 years and 8 months
Population: The Safety Analysis Set included all participants who received ≥ 1 dose of zanubrutinib and/or obinutuzumab. The Safety Analysis Set was the primary analysis set for the efficacy and safety analyses.. Only participants with post-baseline assessments and available data were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1: Zanubrutinib and Obinutuzumab
Number analyzed (Participants) | 22
Months
  Non-GCB DLBCL | 11.93 [3.52 to 16.53]
  CLL/SLL | NA [NA to NA] — NA = Data not estimable due to insufficient number of participants with events
  WM | NA [22.4 to NA] — NA = Data not estimable due to insufficient number of participants with events
  FL | NA [42.45 to NA] — NA = Data not estimable due to insufficient number of participants with events
  MCL | NA [7.92 to NA] — NA = Data not estimable due to insufficient number of participants with events
  MZL | NA [NA to NA] — NA = Data not estimable due to insufficient number of participants with events

11. Secondary Outcome: Part 1 and Part 2: Hematologic Improvement In Participants With CLL
Description: The number and percentage of participants with CLL with anemia (hemoglobin ≤110 grams/liter [g/L]), neutropenia (absolute neutrophil count ≤1.5 x 10^9/L), or thrombocytopenia (platelet count ≤100 x 10^9/L) at baseline were estimated.
Time Frame: Day 1 (first dose) through 4 years and 8 months
Population: The Safety Analysis Set included all participants who received ≥ 1 dose of zanubrutinib and/or obinutuzumab. The Safety Analysis Set was the primary analysis set for the efficacy and safety analyses. Only participants with post-baseline assessments and available data were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Zanubrutinib and Obinutuzumab
Number analyzed (Participants) | 37
Participants
  Participants with anemia at baseline who had normalized hemoglobin after treatment | 11
  Participants with neutropenia at baseline who had normalized hemoglobin after treatment | 3
  Participants with thrombocytopenia at baseline who had normalized hemoglobin after treatment | 12

12. Secondary Outcome: Part 1: Area Under The Plasma Concentration-time Curve From Time 0 To The Time Of The Last Measurable Concentration (AUClast) Of Zanubrutinib
Time Frame: Day 1 Cycle 1, Predose (within 3 hours), hours 1, 2, 4 and 7
Population: The Pharmacokinetic Analysis Set included all participants who received at least the first administration of zanubrutinib and provided PK samples per protocol after the first administration of zanubrutinib on Cycle 1 Day 1. Only participants with available data were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter*hour
Arm/Group | Zanubrutinib and Obinutuzumab
Number analyzed (Participants) | 6
nanogram/milliliter*hour
  160 mg BID | 1123.59 (71.482)
  320 mg QD | 2179.54 (70.237)

13. Secondary Outcome: Part 1: Area Under The Plasma Concentration-time Curve From Time 0 To Infinity Time (AUC) Of Zanubrutinib
Time Frame: Day 1 Cycle 1, Predose (within 3 hours), hours 1, 2, 4 and 7
Population: The PK Analysis Set included all participants who received at least the first administration of zanubrutinib and provided PK samples per protocol (without any significant protocol deviation affecting the PK blood sample) after the first administration of zanubrutinib on Cycle 1 Day 1. Only participants with available data were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter*hour
Arm/Group | Zanubrutinib and Obinutuzumab
Number analyzed (Participants) | 6
nanogram/milliliter*hour
  160 mg BID | 1324.63 (60.981)
  320 mg QD | 3052.47 (33.681)

14. Secondary Outcome: Part 1: Maximum Plasma Concentration (Cmax) Of Zanubrutinib
Time Frame: Day 1 Cycle 1, Predose (within 3 hours), hours 1, 2, 4 and 7
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter
Arm/Group | Zanubrutinib and Obinutuzumab
Number analyzed (Participants) | 6
nanogram/milliliter
  160 mg BID | 360.42 (90.350)
  320 mg QD | 589.37 (79.884)

15. Secondary Outcome: Part 1: Time To Maximum Plasma Concentration (Tmax) Of Zanubrutinib
Time Frame: Day 1 Cycle 1, Predose (within 3 hours), hours 1, 2, 4 and 7
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Zanubrutinib and Obinutuzumab
Number analyzed (Participants) | 6
hour
  160 mg BID | 1.60 (38.285)
  320 mg QD | 1.73 (88.663)

16. Secondary Outcome: Part 1: Terminal Elimination Half-life (t1/2) Of Zanubrutinib
Time Frame: Day 1 Cycle 1, Predose (within 3 hours), hours 1, 2, 4 and 7
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Zanubrutinib and Obinutuzumab
Number analyzed (Participants) | 5
hour
  160 mg BID | 1.88 (29.532)
  320 mg QD | 1.79 (19.945)

17. Secondary Outcome: Part 1: Apparent Clearance (CL/F) Of Zanubrutinib
Time Frame: Day 1 Cycle 1, Predose (within 3 hours), hours 1, 2, 4 and 7
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliter/hour
Arm/Group | Part 1: Zanubrutinib and Obinutuzumab
Number analyzed (Participants) | 5
milliliter/hour
  160 mg BID | 120789.1 (60.965)
  320 mg QD | 104832.9 (33.681)

18. Secondary Outcome: Part 1: Apparent Volume Of Distribution (Vz/F) Of Zanubrutinib
Time Frame: Day 1 Cycle 1, Predose (within 3 hours), hours 1, 2, 4 and 7
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliter
Arm/Group | Part 1: Zanubrutinib and Obinutuzumab
Number analyzed (Participants) | 6
milliliter
  160 mg BID | 327343.8 (97.981)
  320 mg QD: number analyzed (Participants) | 5
  320 mg QD | 270810 (36.099)

19. Secondary Outcome: Part 1 and Part 2: Steady State AUClast Of Zanubrutinib
Time Frame: Day 1 Cycle 1, Predose (within 3 hours), hours 1, 2, 4 and 7
Population: The PK Analysis Set included all participants in Part and Part 2, who received at least the first administration of zanubrutinib and provided PK samples per protocol (without any significant protocol deviation affecting the PK blood sample) after the first administration of zanubrutinib on Cycle 1 Day 1.Only participants with available samples were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter*hour
Arm/Group | Zanubrutinib and Obinutuzumab
Number analyzed (Participants) | 75
nanogram/milliliter*hour
  160 mg BID: number analyzed (Participants) | 36
  160 mg BID | 1074.1 (42.1)
  320 mg QD | 2003.9 (42.6)

20. Secondary Outcome: Part 1 and Part 2: Steady State Cmax of Zanubrutinib
Time Frame: Day 1 Cycle 1, Predose (within 3 hours), hours 1, 2, 4 and 7
Population: The PK Analysis Set included all participants Part and Part 2 who received at least the first administration of zanubrutinib and provided PK samples per protocol (without any significant protocol deviation affecting the PK blood sample) after the first administration of zanubrutinib on Cycle 1 Day 1. Only participants with available data were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter
Arm/Group | Zanubrutinib and Obinutuzumab
Number analyzed (Participants) | 75
nanogram/milliliter
  160 mg BID: number analyzed (Participants) | 36
  160 mg BID | 328.5 (52.3)
  320 mg QD | 580 (42.6)

21. Secondary Outcome: Part 1 and Part 2: Steady State Tmax Of Zanubrutinib
Time Frame: Day 1 Cycle 1, Predose (within 3 hours), hours 1, 2, 4 and 7
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Zanubrutinib and Obinutuzumab
Number analyzed (Participants) | 75
hour
  160 mg BID: number analyzed (Participants) | 36
  160 mg BID | 1.8 (67.0)
  320 mg QD | 1.9 (48.4)

22. Secondary Outcome: Part 2: Number Of Participants Experiencing Adverse Events
Description: An AE was defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product (zanubrutinib in combination with obinutuzumab). An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study drug. An SAE was any untoward medical occurrence that, at any dose,:
  * resulted in death,
  * was life threatening,
  * required hospitalization or prolongation of existing hospitalization,
  * resulted in disability/incapacity,
  * was a congenital anomaly/birth defect.
Time Frame: Day 1 (first dose) through 4 years and 8 months
Population: The Safety Analysis Set included all participants who received ≥ 1 dose of zanubrutinib and/or obinutuzumab.
Measure: Count of Participants; unit: Participants
Groups:
- Part 2: Zanubrutinib and Obinutuzumab: Part 2: The 2 dose regimens selected from Part 1 (zanubrutinib 320 mg QD and 160 mg BID in combination with obinutuzumab) were investigated in 5 expansion cohorts.
Arm/Group | Part 2: Zanubrutinib and Obinutuzumab
Number analyzed (Participants) | 119
Participants
  Any AE | 119
  SAE | 62

23. Secondary Outcome: Part 2: Number Of Participants With Clinical Laboratory Abnormalities
Description: Results are reported as participants with shifts towards (high directionality) or away (low directionality) from Grade 3 or Higher Toxicity.
Time Frame: Day -28 to -1 (predose) through 4 years and 8 months
Population: The Safety Analysis Set included all participants who received ≥ 1 dose of zanubrutinib and/or obinutuzumab. Only participants with available data were included in the analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Part 2: 160 mg BID: Part 2: The 2 dose regimens selected from Part 1 (zanubrutinib 320 mg QD and 160 mg BID in combination with obinutuzumab) were investigated in 5 expansion cohorts.
Arm/Group | Part 2: 160 mg BID
Number analyzed (Participants) | 42
Participants
  Hemoglobin: Low Directionality | 3
  Leukocytes: Low Directionality | 7
  Leukocytes: High Directionality | 0
  Lymphocytes: Low Directionality | 10
  Lymphocytes: High Directionality | 2
  Neutrophils: Low Directionality | 11
  Platelets: Low Directionality | 7
  Alanine Aminotransferase: High Directionality | 1
  Albumin: Low Directionality | 5
  Alkaline Phosphatase: High Directionality | 1
  Aspartate Aminotransferase: High Directionality | 1
  Glucose: High Directionality | 3
  Phosphate: Low Directionality | 3
  Sodium: Low Directionality | 1
  Urate: High Directionality | 1

24. Secondary Outcome: Part 2: Number Of Deaths
Description: An AE was defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product (zanubrutinib in combination with obinutuzumab). An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study drug. An SAE was any untoward medical occurrence that, at any dose,:
  * resulted in death,
  * is life threatening,
  * required hospitalization or prolongation of existing hospitalization,
  * resulted in disability/incapacity,
  * was a congenital anomaly/birth defect.
Time Frame: Day 1 (first dose) through 4 years and 8 months
Population: The Safety Analysis Set included all participants who received ≥ 1 dose of zanubrutinib and/or obinutuzumab
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Zanubrutinib and Obinutuzumab
Number analyzed (Participants) | 119
Participants
  Total deaths | 34
  Progression of disease | 24
  Unknown | 2
  Acute respiratory distress syndrome | 1
  Road traffic accident | 1
  Bone marrow failure and metastatic skin squamous cell carcinoma | 1
  Cardiac arrest during admission to private hospital for bowel resection for colorectal cancer | 1
  Chest infection | 1
  CLL/sepsis | 1
  Metastatic breast cancer | 1
  Undisclosed | 1

ADVERSE EVENTS:
Time Frame: Day 1 (first dose) through 4 years and 8 months
Arm/Group | Zanubrutinib and Obinutuzumab
All-Cause Mortality (participants affected / at risk) | 34/119
Serious Adverse Events (participants affected / at risk) | 62/119
Other Adverse Events (participants affected / at risk) | 119/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zanubrutinib and Obinutuzumab (N=119)
Pneumonia (Infections and infestations) | 8
Influenza (Infections and infestations) | 4
Urinary tract infection (Infections and infestations) | 4
Cellulitis (Infections and infestations) | 3
Gastroenteritis (Infections and infestations) | 3
Sepsis (Infections and infestations) | 3
Appendicitis (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 2
Herpes zoster (Infections and infestations) | 2
Pneumonia pseudomonal (Infections and infestations) | 2
Appendicitis perforated (Infections and infestations) | 1
Campylobacter gastroenteritis (Infections and infestations) | 1
Campylobacter sepsis (Infections and infestations) | 1
Disseminated cryptococcosis (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Gastritis viral (Infections and infestations) | 1
Gastroenteritis aeromonas (Infections and infestations) | 1
Herpes zoster disseminated (Infections and infestations) | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1
Listeriosis (Infections and infestations) | 1
Localised infection (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Lower respiratory tract infection viral (Infections and infestations) | 1
Lung abscess (Infections and infestations) | 1
Picornavirus infection (Infections and infestations) | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1
Pneumonia haemophilus (Infections and infestations) | 1
Pneumonia pneumococcal (Infections and infestations) | 1
Pseudomonal sepsis (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Rhinovirus infection (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Sinusitis bacterial (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Skin squamous cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pyrexia (General disorders) | 8
Multiple organ dysfunction syndrome (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Peripheral swelling (General disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Small intestinal obstruction (Gastrointestinal disorders) | 2
Ascites (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1
Eye contusion (Injury, poisoning and procedural complications) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Hyphaema (Injury, poisoning and procedural complications) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1
Post procedural bile leak (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Sternal fracture (Injury, poisoning and procedural complications) | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1
Neutropenia (Blood and lymphatic system disorders) | 5
Haemolysis (Blood and lymphatic system disorders) | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Haemorrhage intracranial (Nervous system disorders) | 1
Ischaemic stroke (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1
Renal impairment (Renal and urinary disorders) | 2
Haematuria (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1
Confusional state (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 1
Cytokine storm (Immune system disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zanubrutinib and Obinutuzumab (N=119)
Upper respiratory tract infection (Infections and infestations) | 55
Lower respiratory tract infection (Infections and infestations) | 16
Sinusitis (Infections and infestations) | 15
Urinary tract infection (Infections and infestations) | 13
Pneumonia (Infections and infestations) | 12
Bronchitis (Infections and infestations) | 10
Cellulitis (Infections and infestations) | 10
Conjunctivitis (Infections and infestations) | 9
Nasopharyngitis (Infections and infestations) | 9
Herpes zoster (Infections and infestations) | 7
Oral herpes (Infections and infestations) | 6
Gastroenteritis (Infections and infestations) | 4
Onychomycosis (Infections and infestations) | 4
Otitis media (Infections and infestations) | 4
Rash (Skin and subcutaneous tissue disorders) | 23
Petechiae (Skin and subcutaneous tissue disorders) | 18
Night sweats (Skin and subcutaneous tissue disorders) | 9
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 9
Pruritus (Skin and subcutaneous tissue disorders) | 8
Rash erythematous (Skin and subcutaneous tissue disorders) | 8
Dry skin (Skin and subcutaneous tissue disorders) | 5
Skin lesion (Skin and subcutaneous tissue disorders) | 5
Erythema (Skin and subcutaneous tissue disorders) | 4
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 31
Nausea (Gastrointestinal disorders) | 22
Constipation (Gastrointestinal disorders) | 14
Dyspepsia (Gastrointestinal disorders) | 12
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 10
Abdominal pain (Gastrointestinal disorders) | 9
Abdominal distension (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 7
Abdominal pain upper (Gastrointestinal disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 36
Productive cough (Respiratory, thoracic and mediastinal disorders) | 12
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 6
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 5
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 5
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 5
Fatigue (General disorders) | 38
Pyrexia (General disorders) | 18
Oedema peripheral (General disorders) | 15
Chills (General disorders) | 10
Peripheral swelling (General disorders) | 8
Non-cardiac chest pain (General disorders) | 6
Contusion (Injury, poisoning and procedural complications) | 39
Fall (Injury, poisoning and procedural complications) | 10
Skin laceration (Injury, poisoning and procedural complications) | 5
Neutropenia (Blood and lymphatic system disorders) | 41
Thrombocytopenia (Blood and lymphatic system disorders) | 26
Anaemia (Blood and lymphatic system disorders) | 13
Lymphopenia (Blood and lymphatic system disorders) | 6
Increased tendency to bruise (Blood and lymphatic system disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 17
Arthralgia (Musculoskeletal and connective tissue disorders) | 15
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Flank pain (Musculoskeletal and connective tissue disorders) | 5
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4
Dizziness (Nervous system disorders) | 13
Headache (Nervous system disorders) | 13
Peripheral sensory neuropathy (Nervous system disorders) | 8
Lethargy (Nervous system disorders) | 6
Paraesthesia (Nervous system disorders) | 6
Sciatica (Nervous system disorders) | 4
Platelet count decreased (Investigations) | 9
Blood alkaline phosphatase increased (Investigations) | 5
Alanine aminotransferase increased (Investigations) | 4
Blood creatinine increased (Investigations) | 4
Electrocardiogram QT prolonged (Investigations) | 4
Gamma-glutamyltransferase increased (Investigations) | 4
Decreased appetite (Metabolism and nutrition disorders) | 9
Hyperglycaemia (Metabolism and nutrition disorders) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 4
Haematuria (Renal and urinary disorders) | 16
Renal impairment (Renal and urinary disorders) | 5
Proteinuria (Renal and urinary disorders) | 4
Hypertension (Vascular disorders) | 9
Hypotension (Vascular disorders) | 6
Haematoma (Vascular disorders) | 5
Flushing (Vascular disorders) | 4
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7
Vision blurred (Eye disorders) | 5
Insomnia (Psychiatric disorders) | 12
Anxiety (Psychiatric disorders) | 5
Depression (Psychiatric disorders) | 5
Palpitations (Cardiac disorders) | 4
Vertigo (Ear and labyrinth disorders) | 4
Hypogammaglobulinaemia (Immune system disorders) | 8
Seasonal allergy (Immune system disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights.

DOCUMENTS (2):
  • Study Protocol (2019-01-03): https://cdn.clinicaltrials.gov/large-docs/76/NCT02569476/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-03): https://cdn.clinicaltrials.gov/large-docs/76/NCT02569476/SAP_001.pdf